CLINICAL TRIAL: NCT06106048
Title: Comparative Effects of Conscious Abdominal Contraction and Closed Kinetic Chain Exercises on the Activation of Periscapular Muscles in Badminton Players With Subacromial Pain Syndrome
Brief Title: Comparative Effects of Conscious Abdominal Contraction and Closed Kinetic Chain Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCRS &AHS/23/0460
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Subacromial Impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A was treated with closed kinetic chain exercises
  Interventions: Other: Closed kinetic chain exercises
- Group B (Experimental): Group B was treated with abdominal contraction exercises for periscapular activation
  Interventions: Other: Abdominal contraction exercises

INTERVENTIONS:
Other: Closed kinetic chain exercises — Group A was treated with closed kinetic chain exercises. Group A: Group A was treated with closed kinetic chain exercises. Closed kinetic chain exercises enhance the proprioception by coordinating the mechanical receptors as well as the strength of the external shoulder rotator muscles, reduce the pain and improve the shoulder.
  Closed kinetic chain exercises include:
  * Push up
  * Scapular push up
  * Scapular dip
  * Crab walk
  Common Treatment:
  Cryotherapy 10 minutes 2 times per day. Ultrasonography 1Mhz frequency, 0.4 watt/cm for 10 minutes. Transcutaneous electrical stimulation (TENS) 10 minutes, modulation mode, frequency 280, wavelength 80.
  Cross arm stretching 5 times 30 sec hold. Shoulder isometric exercises 10 repetitions 3 sets for 3 times per week.
  Arms: Group A
Other: Abdominal contraction exercises — Group B was treated with abdominal contraction exercises for periscapular activation that includes: Wall slide, knee pushup, external rotation kneeling, Full can and External rotation with elevation and isometric low row.
  Common Treatment:
  Cryotherapy 10 minutes 2 times per day. Ultrasonography 1Mhz frequency, 0.4 watt/cm for 10 minutes. Transcutaneous electrical stimulation (TENS) 10 minutes, modulation mode, frequency 280,wavelength 80.
  Cross arm stretching 5 times 30 sec hold. Shoulder isometric exercises 10 repetitions 3 sets for 3 times per week.
  Arms: Group B

SUMMARY:
Subacromial pain syndrome is a general term used to describe pain which originates from the shoulder and can spread towards the neck or down the arm. It's the most common reason for shoulder pain. The aim of study was to compare the effects of conscious abdominal contraction and closed kinetic chain exercises on the activation of peri-scapular muscles in badminton players with sub-acromial pain syndrome.

DETAILED DESCRIPTION:
A Randomized Clinical Trial was conducted at Sir Syed Sports Complex Sargodha, through convenience sampling technique on 52 patients which was allocated using random sampling through computerized generated number into Group A and Group B. Group A was treated with closed kinetic chain exercises. Group B was treated with abdominal contraction exercises for periscapular activation. These exercises were done in 3 sets with 10 repetitions. There was 3 sessions per week. Baseline measurement was taken on 1st day of evaluation and post treatment will be taken on 4th week. Data was analyzed during SPSS software version 25. After assessing normality of data by Shapiro-Wilk test, it was decided either parametric or non-parametric test was used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Male Badminton players
* Age 20 to 40 years
* Unilateral shoulder pain
* Pain with overhead activities
* Positive Hawkins Kennedy test
* Positive painful arc(60-120 degrees)
* Positive Neer impingement test
* Positive external rotation test
* Numeric pain Rating Scale NPRS value(3-7)

Exclusion Criteria:

* Adhesive capsulitis
* Know shoulder instability
* Neck pain
* Radiating pain from shoulder to hand
* Receiving any intervention for shoulder injury.
* Previous history of 6 month shoulder trauma.
* Previous history of shoulder surgery.
* Taking any critical care medicine

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 28 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-03-23 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
NPRS | upto 4-week
  Patient level of pain will be assessed using this scale. In a Numerical Rating Scale (NRS), this scale ranges from 0 to 10. 0 indicates "no pain" and 10 indicates "worst pain" patients are asked to circle the number between 0 and 10, that fits best to their pain intensity.
  NRS scores ≤ 5 correspond to mild, scores of 6-7 to moderate and scores ≥8 to severe pain in terms of pain-related interference with functioning.
  Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible. The NPRS is a widely used subjective pain measure that has good test-retest reliability (r=. 79-. 96) and validity of NPRS range from 0.86 to 0.95.
SPADI | upto 4-week
  The Shoulder Pain and Disability Index (SPADI) consists of 13 items that have two main domains; in which subscale of 5-item that measures the pain and subscale of 8- item measures disability. The reliability of SPADI ranged from 0.90 to 0.94 and the validity ranged from 0.87 to 0.89.
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.
Universal Goniometer | upto 4-week
  A goniometer will be used in the study to measure shoulder flexion, internal rotation and external rotation.
  Goniometer is an instrument that measures the available range of motion at a joint. To .measure the range of motion physical therapists most commonly use a goniometer. Therapist can use a goniometer to assess what the range of motion is at the initial assessment. The validity of UG (r=0.84 to 0.93) and high intra-rater reliability of goniometer on repeated measures of shoulder range of motions (ICC=0.98-0.99).
Dynamometer | upto 4-week
  A dynamometer will be used in study to measure the strength of serratus anterior muscle, latissimus dorsi muscle, upper and lower trapezius muscles It is is a device that can measure force. The hand-held dynamometer is a small device that fits in the examiner's hand and is placed at precise locations on a subject's limb in an effort to assess the force generated by various muscles or groups of muscles. Inter-tester and intra-tester reliability of digital dynamometer were excellent for all movements (ICC ≥ 0.855) and validity is > 0.913.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Imran Ghafoor, Principal Investigator — Riphah International University
Locations (1):
- Sir Syed Sports Complex, Sargodha, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park SW, Chen YT, Thompson L, Kjoenoe A, Juul-Kristensen B, Cavalheri V, McKenna L. No relationship between the acromiohumeral distance and pain in adults with subacromial pain syndrome: a systematic review and meta-analysis. Sci Rep. 2020 Nov 26;10(1):20611. doi: 10.1038/s41598-020-76704-z. PMID 33244115
- [Background] Saito H, Harrold ME, Cavalheri V, McKenna L. Scapular focused interventions to improve shoulder pain and function in adults with subacromial pain: A systematic review and meta-analysis. Physiother Theory Pract. 2018 Sep;34(9):653-670. doi: 10.1080/09593985.2018.1423656. Epub 2018 Jan 19. PMID 29351510
- [Background] Pieters L, Lewis J, Kuppens K, Jochems J, Bruijstens T, Joossens L, Struyf F. An Update of Systematic Reviews Examining the Effectiveness of Conservative Physical Therapy Interventions for Subacromial Shoulder Pain. J Orthop Sports Phys Ther. 2020 Mar;50(3):131-141. doi: 10.2519/jospt.2020.8498. Epub 2019 Nov 15. PMID 31726927
- [Background] Pogetti LS, Nakagawa TH, Contecote GP, Camargo PR. Core stability, shoulder peak torque and function in throwing athletes with and without shoulder pain. Phys Ther Sport. 2018 Nov;34:36-42. doi: 10.1016/j.ptsp.2018.08.008. Epub 2018 Aug 17. PMID 30145541
- [Background] Overbeek CL, Kolk A, de Groot JH, Visser CPJ, van der Zwaal P, Jens A, Nagels J, Nelissen RGHH. Altered Cocontraction Patterns of Humeral Head Depressors in Patients with Subacromial Pain Syndrome: A Cross-sectional Electromyography Analysis. Clin Orthop Relat Res. 2019 Aug;477(8):1862-1868. doi: 10.1097/CORR.0000000000000745. PMID 31107319
- [Background] de Oliveira Scatolin R, Hotta GH, Cools AM, Custodio GAP, de Oliveira AS. Effect of conscious abdominal contraction on the activation of periscapular muscles in individuals with subacromial pain syndrome. Clin Biomech (Bristol). 2021 Apr;84:105349. doi: 10.1016/j.clinbiomech.2021.105349. Epub 2021 Apr 2. PMID 33848705
- [Background] Silva YA, Novaes WA, Dos Passos MHP, Nascimento VYS, Cavalcante BR, Pitangui ACR, De Araujo RC. Reliability of the Closed Kinetic Chain Upper Extremity Stability Test in young adults. Phys Ther Sport. 2019 Jul;38:17-22. doi: 10.1016/j.ptsp.2019.04.004. Epub 2019 Apr 9. PMID 31035171
- [Background] Cappato de Araujo R, Andrade da Silva H, Pereira Dos Passos MH, Alves de Oliveira VM, Rodarti Pitangui AC. Use of unstable exercises in periscapular muscle activity: A systematic review and meta-analysis of electromyographic studies. J Bodyw Mov Ther. 2021 Apr;26:318-328. doi: 10.1016/j.jbmt.2020.12.010. Epub 2020 Dec 8. PMID 33992265
- [Background] Scott R, Yang HS, James CR, Sawyer SF, Sizer PS Jr. Volitional Preemptive Abdominal Contraction and Upper Extremity Muscle Latencies During D1 Flexion and Scaption Shoulder Exercises. J Athl Train. 2018 Dec;53(12):1181-1189. doi: 10.4085/1062-6050-255-17. Epub 2018 Dec 13. PMID 30543446
- [Background] Werin M, Maenhout A, Smet S, Van Holder L, Cools A. Muscle recruitment during plyometric exercises in overhead athletes with and without shoulder pain. Phys Ther Sport. 2020 May;43:19-26. doi: 10.1016/j.ptsp.2020.01.015. Epub 2020 Feb 1. PMID 32058922